CLINICAL TRIAL: NCT05331469
Title: Difference of Basal Insulin Titration Method in Reducing HbA1c Among Type 2 Diabetes Mellitus (T2DM) Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021525-10165
Record Dates: First submitted 2022-04-11; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: to Identify Which Titration Regimen of Basal Insulin (Being Daily Titration vs 3 Daily Titration) is Better in Reducing hba1c and Have Lesser Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily basal insulin titration (Active Comparator): Participants in this intervention arm will be started with basal insulin of 10 units or 0.2 unit/kg (whichever lower) at pre-bed time. They will then check their morning fasting CBG the following day. If they have no hypoglycemia symptoms or documented hypoglycemic CBG (<3.9mmol/L), and their fasting CBG is more than 7mmol/L, they will then self-titrate their basal insulin by 1 unit (ie 10+1) the following night. This same process is going to be repeated until their fasting CBG achieve 7mmol/L or lower. Then, they will continue and maintain on the desired basal insulin dosage till their appointment. The maximum basal insulin that is allowed to be titrated by the participants is up to 0.5unit/kg. Participants are required to document down their CBG and any hypoglycemia symptoms in a simple table method provided to them
  Interventions: Drug: NPH basal insulin titration
- 3 daily basal insulin titration (Active Comparator): Participants in this intervention arm will be started with basal insulin of 10 units or 0.2 unit/kg (whichever lower) at pre-bed time. They will then check their morning fasting CBG the following 3 days. If they have no hypoglycemia symptoms or documented hypoglycemic CBG (<3.9mmol/L), and their fasting CBG is more than 7mmol/L (for 2 out of 3 days), they will then self-titrate their basal insulin by 2 units (ie 10+2) on the 3rd night. This same process is going to be repeated until their fasting CBG achieved 7mmol/L or lower. Then, they will continue and maintain on the desired basal insulin dosage till their appointment. The maximum basal insulin that is allowed to be titrated by the participants is up to 0.5unit/kg. Participants are required to document down their CBG and any hypoglycemia symptoms in a simple table method provided to them.
  Interventions: Drug: NPH basal insulin titration

INTERVENTIONS:
Drug: NPH basal insulin titration — Comparing both arms NPH basal insulin titration in reducing hba1c after 3 months

SUMMARY:
Introduction Diabetes mellitus is a worrying global non-communicable disease where it is affecting 18.3% of Malaysian adults. Poorly managed diabetes leads to an array of serious complications, namely heart attack, kidney failure and stroke. Insulin therapy remains one of the most important medication in treating diabetes especially in the population with high sugar readings or long standing diabetes. Outpatient consultations for T2DM patients are spaced out due to the limited amount of treating physicians and clinic time. This resorts to the importance of outpatient patient-lead insulin titration. Different guidelines from local and international showed different basal insulin titration method in achieving ideal fasting blood sugar.

Objective We aim to investigate the difference of basal insulin titration methods in reducing HbA1c among the T2DM patients.

Methodology In a parallel group randomized controlled trial, we aim to recruit 70 adult T2DM patients who have poorly controlled T2DM ( HbA1c > 7.5% with FPG >8mmol/L) or newly diagnosed T2DM patients (who are symptomatic or HbA1c >10% or FPG >13 mmol/L). The subjects will be randomized to 2 groups, daily basal insulin titration and 3 daily basal insulin titration. These subjects will be follow up for 12 weeks (4th week and 8th week virtual consultation and 12th week face-to-face consultation). The primary outcome is the HbA1c reduction from baseline to the end of 12weeks intervention. The secondary outcomes are percentage of T2DM patients achieving fasting blood sugar within 4.4-7mmol/L and/or HbA1c <7% within the study period, the incidence of hypoglycemia, total daily basal insulin dosage required to achieve desired fasting blood sugar, duration taken to achieve desired fasting blood sugar, weight changes and satisfaction to the therapy between the 2 intervention groups.

Clinical Significance This study enables us to evaluate the efficacy of the different basal insulin titration methods among the T2DM patients.

DETAILED DESCRIPTION:
Hypothesis Daily basal insulin titration reduces HbA1c more significantly compared with 3 daily basal insulin titration among T2DM patients.

Aims

Primary Aim :

To evaluate the difference of daily basal insulin titration method and 3-daily basal insulin titration method in reducing HbA1c among T2DM patients

Secondary Aim :

To evaluate the percentage of T2DM patients achieving fasting blood sugar within 4.4-7mmol/L and/or HbA1c below 7% within the study period, frequency of hypoglycemia, total daily basal insulin dosage needed to achieve fasting capillary blood glucose 4.4-7mmol/L, duration taken to achieve optimal fasting capillary blood glucose 4.4-7mmol/L, weight changes and satisfaction to the titration therapy between the daily basal insulin and 3-daily basal insulin titration method.

Background and Clinical Significance Background Diabetes Mellitus is a worrying non communicable disease both locally and globally. Malaysia Nasional Heath and Morbidity Survey 2019 (NHMS 2019) reported the prevalence of diabetes mellitus was 18.3%, an increase from year 2011 (11.2%) and year 2015 (13.4%). With the prevalence of nearing 1 in 5 adult Malaysian suffering from diabetes mellitus, a good control of the disease is the ultimate way to prevent diabetes related complications from occurring, namely stroke, heart attack and kidney failure.

Insulin is one of the most widely used injectable diabetic medications that is suitable to be incorporated with a wide range of antidiabetic medications such as oral antidiabetic drugs (OAD) and GLP-1 receptor agonists (GLP-1 RA). Insulin therapy should be considered in T2DM patients that have inadequate glycemic control (HbA1c >7.5% with Fasting capillary blood glucose (CBG) >8 mmol/L) on optimal OADs and it should also be used as an initial therapy in newly diagnosed T2DM patients who are symptomatic (osmotic symptoms), Hba1c >10% or fasting plasma glucose >13mmol/L.

The enormous diabetic patients in Malaysia, largely managed in governmental clinic/ hospital setting pose the technical difficulty for clinicians to review them at regular basis. An average duration of a face-to-face consultation at an outpatient setting is scheduled at 3 monthly to 6 monthly intervals. This makes it a technical difficulty for insulin users to titrate their medications if they are purely managed by clinicians. Patient-lead basal insulin titration has been proven to be more effective than clinician-driven insulin titration to achieve the HbA1c target. It is also proven that outpatient patient-lead basal insulin titration is easy to achieve targeted HbA1c compared with clinician-driven OADs titration.

Local Malaysia CPG guideline suggested weekly basal insulin titration to achieve glycemic target.2 Where else American Diabetes Association 2019 advocate adjustment of basal insulin by 2-4 units once or twice a week to achieve the desired fasting blood sugar level.6 In the context of Canadian 2018 Diabetes CPG, they suggest 1 unit daily adjustment of basal insulin to achieve targeted fasting blood sugar level.7 Various studies using different patient-lead basal insulin titration regimen ranging from 1 unit per day to 2-3 units every 3 days have proven to be efficacious and safe in achieving HbA1c target among the T2DM patients.

Clinical Significance This study hopes to achieve a best outpatient patient-lead basal insulin titration whether daily 1 unit titration or 3 daily 2 units titration is better in achieving the targeted HbA1c. This will also enable us to evaluate which titration regimen is safer and easier to adhere among T2DM patients who require basal insulin commencement.

Study Design This study is designed as a parallel group randomized controlled trial with 12 weeks of intervention and follow up. The total duration of participation is 12 weeks.

Participants Adult T2DM patients Inclusion Criteria

1. Adults aged 18 years and above
2. HbA1c >7.5% and Fasting blood sugar > 8mmol/L
3. Newly diagnosed T2DM with osmotic symptoms or HbA1c >10% or FPG >13mmol/L
4. Insulin naïve patients
5. Patients planned for insulin initiation
6. Ability to give informed consent
7. Ability to perform self-monitoring blood glucose

Exclusion Criteria

1. Diabetes other than type 2 diabetes mellitus
2. Diabetes in pregnancy
3. Diabetes with chronic kidney disease stage 3,4 and 5 (eGFR <60ml/min/1.73m2)
4. Patient with history of severe hypoglycemia
5. Active proliferative diabetic retinopathy
6. Any medical condition that may influence HbA1c measurements (e.g., thalassemia, sickle cell anemia)
7. Treatment with systemic corticosteroid

Intervention Basal insulin daily titration arm Participants in this intervention arm will be started with basal insulin of 10 units or 0.2 unit/kg (whichever lower) at pre-bed time. They will then check their morning fasting CBG the following day. If they have no hypoglycemia symptoms or documented hypoglycemic CBG (<3.9mmol/L), and their fasting CBG is more than 7mmol/L, they will then self-titrate their basal insulin by 1 unit (ie 10+1) the following night. This same process is going to be repeated until their fasting CBG achieve 7mmol/L or lower. Then, they will continue and maintain on the desired basal insulin dosage till their appointment. The maximum basal insulin that is allowed to be titrated by the participants is up to 0.5unit/kg. Participants are required to document down their CBG and any hypoglycemia symptoms in a simple table method provided to them.

At any instance if their morning fasting CBG is higher than 14mmol/L, phone consultation can be made to the investigator and further titration of medication or further plans will be instructed by the investigator. If their overnight CBG is <3.9mmol/L, participants are instructed to reduce their basal insulin by 10-20%. Participants are able to contact the investigator if they experience hypoglycemic symptoms if they are unsure of the subsequent steps.

A clear hypoglycemia action plan will be provided to all participants.

Basal insulin 3-daily titration arm Participants in this intervention arm will be started with basal insulin of 10 units or 0.2 unit/kg (whichever lower) at pre-bed time. They will then check their morning fasting CBG the following 3 days. If they have no hypoglycemia symptoms or documented hypoglycemic CBG (<3.9mmol/L), and their fasting CBG is more than 7mmol/L (for 2 out of 3 days), they will then self-titrate their basal insulin by 2 units (ie 10+2) on the 3rd night. This same process is going to be repeated until their fasting CBG achieved 7mmol/L or lower. Then, they will continue and maintain on the desired basal insulin dosage till their appointment. The maximum basal insulin that is allowed to be titrated by the participants is up to 0.5unit/kg. Participants are required to document down their CBG and any hypoglycemia symptoms in a simple table method provided to them.

At any instance if their morning CBG is higher than 14mmol/L, phone consultation can be made to the investigator and further titration of medication or further plans will be instructed by the investigator. If their overnight CBG is <3.9mmol/L, participants are instructed to reduce their basal insulin by 10-20%. Participants are able to contact the investigator if they experience hypoglycemic symptoms if they are unsure of the subsequent steps.

A clear hypoglycemia action plan will be provided to all participants.

Hypoglycemia, Classification and Action Plans Hypoglycemia is defined by either - CBG <3.9mmol/L - Presence of autonomic or neuroglycopenic symptoms - Reversed by carbohydrate (CHO) intake Classification Level 1 - CBG 3-3.9mmol/L Level 2 - CBG <3mmol/L Level 3 - Hypoglycemia requires assistance from another person for recovery

Action Plans Level 1 & 2

* consume 15g of CHO (eg: 1 tablespoon of honey, 150-200ml of fruit juice or soft drink or 3 teaspoons of table sugar dissolve in water)
* repeat CBG within 15 minutes
* if CBG is still < 3.9mmol/L, consume another 15g of CHO (to be repeated until CBG>3.9mmol/L) - if CBG is >3.9mmol/L, to reduce basal insulin by 10-20%

Level 3 - if patient is still conscious, follow steps for Level 1 & 2 - if patient is unconscious, to rush to emergency department

Outcomes measures

1. Primary Outcome

   a. To compare the HbA1c reduction of the daily basal insulin titration arm with the 3-daily basal insulin titration arm
2. Secondary Outcome

   1. To compare the percentage of patient achieving fasting blood glucose within 4.4-7mmol/L and/or HbA1c below 7% between the daily basal insulin titration arm with the 3-daily basal insulin titration arm within the study period
   2. To compare the frequency of hypoglycemia between the daily basal insulin titration arm with the 3- daily basal insulin titration arm
   3. To compare the total basal insulin dosage required to achieve normal fasting CBG 4.4-7.0mmol/L between the daily basal insulin titration arm with the 3-daily basal insulin titration arm
   4. To compare the duration taken to achieve normal fasting CBG 4.4-7.0mmol/L between the daily basal insulin titration arm with the 3-daily basal insulin titration arm
   5. To compare the satisfaction to the titration method between the daily basal insulin titration arm with the 3-daily basal insulin titration arm
   6. To compare with weight changed between the daily basal insulin titration arm with the 3-daily basal insulin titration arm

Study Protocol Week 0 Upon enrolment, demographic data will be collected. Fasting plasma glucose and HbA1c records will be collected. Both intervention groups will receive glucometer devices and strips; they will be advised to record their CBG readings and the hypoglycemic symptoms on the tables given.

Week 4 and Week 8 Teleconsultation will be made by the investigator to ensure the optimal dosages of basal insulins are commenced. Any doubts and difficulties along the titration will be answered during the teleconsultations.

Week 12 Face-to-face consultation will be made. Blood taking will be collected for HbA1c and FPG during the visit. Handling of the recorded glucose-reading table will be done. A simple questionnaire regarding satisfaction of the titration regimen will be carried out. Participants will be discharged back to their previous physician care.

Data analysis and interpretation

Patients' demographic and clinical characteristics at baseline will be compared between the intervention arm 1 and intervention arm 2. Continuous data will be summarized as means (±standard deviation) and categorical data will be summarized as frequencies (%). Depending on the normality distribution, continuous outcomes will be compared between those in the arm 1 and arm 2 groups using a two-sample t-test or Mann-Whitney U test while categorical outcomes will be compared using the Fisher's exact test or Chi-square test. The treatment effect will be expressed as relative risk (95% CI). A p value of <0.05 will be considered significant.

5. Sample Size Calculation Anticipating 10% dropout from each group, A total of (32+32) X 1.1 = 70 subjects will be recruited in the study Mean HbA1c for 3 daily basal insulin adjustment is 7.8% [AT.LANTUS] Mean HbA1c for daily basal insulin adjustment is 6.96% [Canadian INSIGHT]

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus patients with

  1. Adults aged 18 years and above
  2. HbA1c >7.5% and Fasting blood sugar > 8mmol/L
  3. Newly diagnosed T2DM with osmotic symptoms or HbA1c >10% or FPG >13mmol/L
  4. Insulin naïve patients
  5. Patients planned for insulin initiation
  6. Ability to give informed consent
  7. Ability to perform self-monitoring blood glucose

Exclusion Criteria:

1. Diabetes other than type 2 diabetes mellitus
2. Diabetes in pregnancy
3. Diabetes with chronic kidney disease stage 3,4 and 5 (eGFR <60ml/min/1.73m2)
4. Patient with history of severe hypoglycemia
5. Active proliferative diabetic retinopathy
6. Any medical condition that may influence HbA1c measurements (e.g., thalassemia, sickle cell anemia)
7. Treatment with systemic corticosteroid

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Hba1c reduction | 3 months
  To compare the HbA1c reduction of the daily basal insulin titration arm with the 3-daily basal insulin titration arm

SECONDARY OUTCOMES:
percentage of subjects achieving fasting capillary blood glucose and/or hba1c below 7% | 3 months
  To compare the percentage of patient achieving fasting blood glucose within 4.4-7mmol/L and/or HbA1c below 7% between the daily basal insulin titration arm with the 3-daily basal insulin titration arm within the study period
Hypoglycemia frequency | 3 months
  To compare the frequency of hypoglycemia between the daily basal insulin titration arm with the 3- daily basal insulin titration arm
Basal insulin required to achieve fasting blood sugar less than 7mmol/L | 3 months
  To compare the total basal insulin dosage required to achieve normal fasting CBG 4.4-7.0mmol/L between the daily basal insulin titration arm with the 3-daily basal insulin titration arm
Duration to achieve fasting cappilary blood glucose less than 7mmol/L | 3 months
  To compare the duration taken to achieve normal fasting CBG 4.4-7.0mmol/L between the daily basal insulin titration arm with the 3-daily basal insulin titration arm
Satisfaction of titration | 3 months
  To compare the satisfaction to the titration method between the daily basal insulin titration arm with the 3-daily basal insulin titration arm
Weight changes after intervention | 3 months
  To compare with weight changed between the daily basal insulin titration arm with the 3-daily basal insulin titration arm

CONTACTS AND LOCATIONS:
Overall Officials: Yi Jiang Chua, Study Chair — Universiti Malaya Medical Centre
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davies M, Storms F, Shutler S, Bianchi-Biscay M, Gomis R; ATLANTUS Study Group. Improvement of glycemic control in subjects with poorly controlled type 2 diabetes: comparison of two treatment algorithms using insulin glargine. Diabetes Care. 2005 Jun;28(6):1282-8. doi: 10.2337/diacare.28.6.1282. PMID 15920040
- [Background] Davies M, Bain S, Charpentier G, Flacke F, Goyeau H, Woloschak M, Hasslacher C, Vespasiani G, Edelman S. A Randomized Controlled, Treat-to-Target Study Evaluating the Efficacy and Safety of Insulin Glargine 300 U/mL (Gla-300) Administered Using Either Device-Supported or Routine Titration in People With Type 2 Diabetes. J Diabetes Sci Technol. 2019 Sep;13(5):881-889. doi: 10.1177/1932296818821706. Epub 2019 Jan 15. PMID 30646755
- [Background] Gerstein HC, Yale JF, Harris SB, Issa M, Stewart JA, Dempsey E. A randomized trial of adding insulin glargine vs. avoidance of insulin in people with Type 2 diabetes on either no oral glucose-lowering agents or submaximal doses of metformin and/or sulphonylureas. The Canadian INSIGHT (Implementing New Strategies with Insulin Glargine for Hyperglycaemia Treatment) Study. Diabet Med. 2006 Jul;23(7):736-42. doi: 10.1111/j.1464-5491.2006.01881.x. PMID 16842477
- [Background] American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S90-S102. doi: 10.2337/dc19-S009. PMID 30559235
- [Background] Meneghini L, Koenen C, Weng W, Selam JL. The usage of a simplified self-titration dosing guideline (303 Algorithm) for insulin detemir in patients with type 2 diabetes--results of the randomized, controlled PREDICTIVE 303 study. Diabetes Obes Metab. 2007 Nov;9(6):902-13. doi: 10.1111/j.1463-1326.2007.00804.x. PMID 17924873